CLINICAL TRIAL: NCT05865873
Title: Improving Maternal Health Service Utilization Among Women of Reproductive Age in Sidama Regional State, Ethiopia
Brief Title: Maternal Health Service Utilization Among Women of Reproductive Age in Sidama Region, Ethiopia
Acronym: MHSU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hawassa University (Other)
Collaborators: Universidad Pública de Navarra (Other)
Responsible Party: Principal Investigator, Amanuel Yoseph Samago, Lecturer, Hawassa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB/076/15
Record Dates: First submitted 2023-04-03; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Maternal Death
Keywords: Health education, maternal health, utilization, Ethiopia.
MeSH Terms: conditions — Maternal Death; Health Education; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Parallel-group Cluster Randomized Controlled Trial (CRCT) will be used to address the objectives of the current study. The study is a 2 arm CRCT, with every cluster being kebeles located in the Dale and Wonsho districts of Sidama region, Ethiopia. The hallmark of this design is each cluster remains in the arm it was randomly assigned to during the course of the whole study period. Thus, all study subjects are randomly assigned into a group and all the study subjects in the assigned group obtain or do not obtain an intervention.
Who Masked: Outcomes Assessor
Masking Description: Because of the nature of the study intervention, neither research team members nor study respondents can be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Intervention group: will receive routine plus pre-recorded audio-based HEI package for six months until date of delivery.
  Interventions: Behavioral: Health education
- Comparator group (Active Comparator): Comparator group: will receive the routine health education package for six months until the date of delivery as per the Ethiopian guidelines.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Health education — Health education will be delivered for six months, two times per month; one session will take one hour, and an overall 12 sessions will be conducted. One health education session consists of key messages on normal pregnancy and childbirths, ODS during pregnancy, delivery, and the postpartum period, the practice of BPCR, and the benefits of MHSU. The other actions executed by WDT facilitators will be the motivating mother and their families to utilize MHS. One hour will be allocated for each session, from this 20 minutes will be allowed for the pre-recorded an audio-based lecturer and the remaining 40 minutes will be allowed for raising questions and responses (discussion). After the session, some of the women will be selected to carry out role play which is basic to demonstrate the important messages and share experiences.

SUMMARY:
Introduction: Maternal health service (MHS) utilization helps to decrease maternal morbidity and mortality. However, the existing evidence is not sufficient to design effective and efficient strategies.

Objective: This study aims to improve maternal health service utilization among women of reproductive age in the Dale and Wonsho districts of the Sidama region, Ethiopia.

Methods: A community-based cross-sectional study will be carried out to assess the utilization and predictors of maternal health care. A phenomenological qualitative study will be conducted to explore perceptions, barriers, and facilitators of maternal health care. A cluster randomized controlled trial will be employed to assess the effect of health education on maternal knowledge about obstetric danger signs, birth preparedness and complication readiness plan, and maternal health service utilization (MHSU). The minimum required sample size is 1,104 for a cross-sectional study. To explore perceptions, barriers, and facilitators of maternal health care a minimum of 20 in-depth interviews, 3 focus group discussions per group, and 20 key informative interviews will be conducted. The minimum required sample size to assess the effect of health education on outcomes is 942. Data will be entered into Epi Data version 3.1 and exported to the SPSS and Stata software for analysis. Descriptive analyses will be carried out to get descriptive measures for the important variables of interest. The generalized estimated equations analysis will be used to assess the potential predictors of MHSU. The coding and analysis of the qualitative data will be done using the thematic content analysis technique by Atlas-Ti software and presented in narratives.

Schedule and budget: This study will be conducted from October to August 2023; the total cost of the project will be 421,600 ETB (7,026.67 EURO).

DETAILED DESCRIPTION:
Introduction: Maternal health service (MHS) utilization helps to decrease maternal morbidity and mortality. However, the utilization of MHS is low in Ethiopia compared to the national target and is a complex phenomenon affected by several predictors. Its predictors, barriers, and facilitators differ from region to region in Ethiopia, and existing evidence is not adequate to design effective and efficient intervention strategies. One of the methods to increase the utilization of maternal health care is improving maternal knowledge about obstetric danger signs, skills of birth preparedness, and complication readiness practice using health education. However, the effect of health education on these outcomes had not been comprehensively explored and the presently existing studies reported controversial results.

Objective: This study aims to improve maternal health service utilization among women of reproductive age in the North Zone of the Sidama region, Ethiopia.

Methods: A community-based cross-sectional study will be carried out to assess the utilization and predictors of maternal health care. A phenomenological qualitative study will be conducted to explore perceptions, barriers, and facilitators of maternal health care. A cluster randomized controlled trial will be employed to assess the effect of health education on maternal knowledge about obstetric danger signs, birth preparedness and complication readiness plan, and maternal health service utilization. The minimum required sample size is 1,104 for a cross-sectional study. To explore perceptions, barriers, and facilitators of maternal health care a minimum of 20 in-depth interviews, 3 focus group discussions per group, and 20 key informative interviews will be conducted. The minimum required sample size is 942 for the interventional study. A multi-stage sampling method will be used to select the study participants for a cross-sectional study. A maximum variance sampling method will be used for the qualitative study. A cluster-randomized sampling method will be utilized for the interventional study. Quantitative data will be collected using a validated, pre-tested, and structured questionnaire. Qualitative data will be collected using pre-tested focus group discussions, in-depth interviews, and key informant interview guides until information saturation is reached. The intervention group will be received 12 rounds of pre-recorded audio-based health education. The utilization of maternal health care will be measured at baseline and 6 months after the intervention. Data will be entered into Epi Data version 3.1 and exported to the SPSS and Stata software for analysis. Descriptive analyses will be carried out to get descriptive measures for the important variables of interest. The generalized estimated equations (GEE) analysis will be used to assess the potential predictors of MHSU. The coding and analysis of the qualitative data will be done using the thematic content analysis technique by Atlas-Ti software and presented in narratives. For maternal knowledge about the danger signs and practice of birth preparedness and complication readiness, the multilevel linear regression models will be utilized. The generalized mixed models or GEE will be utilized to adjust for between and within-cluster variation for MHSU. The intention-to-treat analysis will be used to compare outcomes between groups. The independent t-tests will be used to compare the effect of the intervention between the two groups. The statistical significance level will be adjusted to account for the effect of multiple comparison problems using the Bonferroni corrections methods.

Schedule and budget: This study will be conducted from December 2022 to December 2023; the total cost of the project will be 421,600 ETB (7,026.67 EURO) and funded by Hawassa University and the Sidama Regional State Administration.

ELIGIBILITY:
Inclusion Criteria

* All pregnant mothers residing in the selected kebeles for at least for 6 months.
* Must haven't planned to change residence during the implementation of an intervention
* No psychiatric problems
* Capable of providing written informed consent
* Voluntary to be visited by WDT facilitators, data collectors, and supervisors. Exclusion Criteria
* Women who have a severe illness during the data collection period.
* Women who experienced stillbirth and infant deaths.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Women of reproductive age
Enrollment: 1126 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of health education intervention on maternal health service utilization among women of reproductive age in North Zone of the Sidama region, Ethiopia. | 6 months
  After the end of intervention period the maternal health service utilization will be measure using the yes and no responses by women's self report
To assess the effect of health education intervention on the knowledge of mothers regarding obstetric danger signs and birth preparedness and complication reediness practice among women of reproductive age in North Zone of the Sidama region, Ethiopia. | 6 months
  After the end of intervention period the obstetric danger signs and birth preparedness and complication readiness will be measure using the yes and no responses by women's self report

CONTACTS AND LOCATIONS:
Overall Officials: Amanuel Samago, Principal Investigator — HAWASSA UNIVERSITY COLLEGE OF MEDICINE AND HEALTH SCIENCES
Locations (1):
- Hawassa University College of Medicine and Health Sciences, Awasa, Sidama Region, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
The findings of the study will be published in peer-reviewed international journals and discussed at national and international seminars and scientific conferences. Also, the findings will be officially presented to the Hawassa University School of Public Health. The summary of the main findings will be delivered to the district health office and the Sidama region health bureau. The findings will also be distributed to vital stakeholders in maternal health policy, comprising the WHO.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 09/08/2024
Access Criteria: un on request from primary author

REFERENCES:
- [Background] Central Statistical Agency (CSA). "[Ethiopia] and ICF," Ethiopia Minin Demographic and Health Survey 2019: Key Indicators Report: Addis Ababa, Ethiopia, and Rockville, CSA and ICF, Maryland, USA.
- [Background] Umar NJ, Afolayan JL, Emmanuel EA, Rejuaro FM, Onasoga OA, et al. (2017) Impact of Health Education on Knowledge and Access to Delivery Care Services by Women among Edu Local Government Area, Nigeria. J Community Med Health Educ 7: 510. doi:10.4172/2161-0711.1000510
- [Background] UM Ango, MO Oche, IS Abubakar, KJ Awosan, Kaoje AU, MO Raji. Effect of health education intervention on knowledge and utilization of health facility delivery services by pregnant women in Sokoto State, Nigeria. International Journal of Contemporary Medical Research 2018;5(6):F4-F9.
- [Background] Jibril UN, Saleh GN, Kayode OS, Morisola RF, Umar A, et al. Impact of Health Education Intervention on Knowledge and Utilization of Postnatal Care Services among Women in Edu Local Government of Kwara State, Nigeria doi: 10.4103/2278-960X.194496
- [Background] OKAFOR, Orji Urenna; YEWANDE, Ademuyiwa Iyabo. Effect of antenatal education on knowledge and utilization of facility-based delivery services among pregnant women in two health institutions in Alimosho, Lagos state. International Journal of Research in Medical Sciences, [S.l.], v. 8, n. 10, p. 3457-3462, sep. 2020. ISSN 2320-6012.
- [Background] Creswell J. W, Qualitative Inquiry & Research Design: Choosing Among Five Traditions. Thousand Oaks: CA. Sag Publications, Inc. 1998.
- [Result] World Health Organization (WHO), Maternal mortality. Available from https://www.who.int/news-room/fact-sheets/detail/maternal-mortality
- [Result] Borde MT, Loha E, Johansson KA, Lindtjorn B. Utilisation of health services fails to meet the needs of pregnancy-related illnesses in rural southern Ethiopia: A prospective cohort study. PLoS One. 2019 Dec 4;14(12):e0215195. doi: 10.1371/journal.pone.0215195. eCollection 2019. PMID 31800574
- [Result] Borde MT, Loha E, Johansson KA, Lindtjorn B. Financial risk of seeking maternal and neonatal healthcare in southern Ethiopia: a cohort study of rural households. Int J Equity Health. 2020 May 18;19(1):69. doi: 10.1186/s12939-020-01183-7. PMID 32423409
- [Result] Borde MT, Loha E, Lindtjorn B. Incidence of postpartum and neonatal illnesses and utilization of healthcare services in rural communities in southern Ethiopia: A prospective cohort study. PLoS One. 2020 Aug 27;15(8):e0237852. doi: 10.1371/journal.pone.0237852. eCollection 2020. PMID 32853242
- [Result] Abosse Z, Woldie M, Ololo S. Factors influencing antenatal care service utilization in hadiya zone. Ethiop J Health Sci. 2010 Jul;20(2):75-82. doi: 10.4314/ejhs.v20i2.69432. PMID 22434964
- [Result] Mamuye SA. Magnitude and Determinants of Postnatal Care Service Utilization Among Women Who Gave Birth in the Last 12 Months in Northern Ethiopia: A Cross-Sectional Study. Int J Womens Health. 2020 Nov 13;12:1057-1064. doi: 10.2147/IJWH.S269704. eCollection 2020. PMID 33223856
- [Result] Geleto A, Chojenta C, Taddele T, Loxton D. Association between maternal mortality and caesarean section in Ethiopia: a national cross-sectional study. BMC Pregnancy Childbirth. 2020 Oct 6;20(1):588. doi: 10.1186/s12884-020-03276-1. PMID 33023536
- [Result] Berelie Y, Yeshiwas D, Yismaw L, Alene M. Determinants of institutional delivery service utilization in Ethiopia: a population based cross sectional study. BMC Public Health. 2020 Jul 8;20(1):1077. doi: 10.1186/s12889-020-09125-2. PMID 32641020
- [Result] Kifle D, Azale T, Gelaw YA, Melsew YA. Maternal health care service seeking behaviors and associated factors among women in rural Haramaya District, Eastern Ethiopia: a triangulated community-based cross-sectional study. Reprod Health. 2017 Jan 13;14(1):6. doi: 10.1186/s12978-016-0270-5. PMID 28086926
- [Result] Ayalew TW, Nigatu AM. Focused antenatal care utilization and associated factors in Debre Tabor Town, northwest Ethiopia, 2017. BMC Res Notes. 2018 Nov 16;11(1):819. doi: 10.1186/s13104-018-3928-y. PMID 30445991
- [Result] Aktac S, Sabuncular G, Kargin D, Gunes FE. Evaluation of Nutrition Knowledge of Pregnant Women before and after Nutrition Education according to Sociodemographic Characteristics. Ecol Food Nutr. 2018 Nov-Dec;57(6):441-455. doi: 10.1080/03670244.2018.1544561. Epub 2018 Nov 13. PMID 30421984
- [Result] Masoi TJ, Kibusi SM. Improving pregnant women's knowledge on danger signs and birth preparedness practices using an interactive mobile messaging alert system in Dodoma region, Tanzania: a controlled quasi experimental study. Reprod Health. 2019 Dec 12;16(1):177. doi: 10.1186/s12978-019-0838-y. PMID 31831076
- [Result] Fetohy EM. Impact of a simple health education program about antenatal care on knowledge, attitudes, subjective norms and intention of pregnant women. J Egypt Public Health Assoc. 2004;79(3-4):283-310. PMID 16918151
- [Result] Kamau M, Mirie W, Kimani S, Mugoya I. Effect of community based health education on knowledge and attitude towards iron and folic acid supplementation among pregnant women in Kiambu County, Kenya: A quasi experimental study. PLoS One. 2019 Nov 25;14(11):e0224361. doi: 10.1371/journal.pone.0224361. eCollection 2019. PMID 31765422
- [Result] Vural F, Vural B. The effect of prenatal and postnatal education on exclusive breastfeeding rates. Minerva Pediatr. 2017 Feb;69(1):22-29. doi: 10.23736/S0026-4946.16.04183-9. PMID 28102653
- [Result] Caine VA, Smith M, Beasley Y, Brown HL. The impact of prenatal education on behavioral changes toward breast feeding and smoking cessation in a healthy start population. J Natl Med Assoc. 2012 May-Jun;104(5-6):258-64. doi: 10.1016/s0027-9684(15)30159-0. PMID 22973675
- [Result] Lassi ZS, Kedzior SG, Bhutta ZA. Community-based maternal and newborn educational care packages for improving neonatal health and survival in low- and middle-income countries. Cochrane Database Syst Rev. 2019 Nov 5;2019(11):CD007647. doi: 10.1002/14651858.CD007647.pub2. PMID 31686427
- [Result] Shimpuku Y, Madeni FE, Horiuchi S, Kubota K, Leshabari SC. A family-oriented antenatal education program to improve birth preparedness and maternal-infant birth outcomes: A cross sectional evaluation study. Reprod Health. 2019 Jul 16;16(1):107. doi: 10.1186/s12978-019-0776-8. PMID 31311563
- [Result] Izudi J, Akwang DG, McCoy SI, Bajunirwe F, Kadengye DT. Effect of health education on birth preparedness and complication readiness on the use of maternal health services: A propensity score-matched analysis. Midwifery. 2019 Nov;78:78-84. doi: 10.1016/j.midw.2019.08.003. Epub 2019 Aug 5. PMID 31400596
- [Result] Soriano-Vidal FJ, Vila-Candel R, Soriano-Martin PJ, Tejedor-Tornero A, Castro-Sanchez E. The effect of prenatal education classes on the birth expectations of Spanish women. Midwifery. 2018 May;60:41-47. doi: 10.1016/j.midw.2018.02.002. Epub 2018 Feb 8. PMID 29486388
- [Result] Bolam A, Manandhar DS, Shrestha P, Ellis M, Costello AM. The effects of postnatal health education for mothers on infant care and family planning practices in Nepal: a randomised controlled trial. BMJ. 1998 Mar 14;316(7134):805-11. doi: 10.1136/bmj.316.7134.805. PMID 9549449
- [Result] Belizan JM, Barros F, Langer A, Farnot U, Victora C, Villar J. Impact of health education during pregnancy on behavior and utilization of health resources. Latin American Network for Perinatal and Reproductive Research. Am J Obstet Gynecol. 1995 Sep;173(3 Pt 1):894-9. doi: 10.1016/0002-9378(95)90362-3. PMID 7573265
- [Result] MacArthur C, Jolly K, Ingram L, Freemantle N, Dennis CL, Hamburger R, Brown J, Chambers J, Khan K. Antenatal peer support workers and initiation of breast feeding: cluster randomised controlled trial. BMJ. 2009 Jan 30;338:b131. doi: 10.1136/bmj.b131. PMID 19181730
- [Result] Central Statistical Agency (CSA) [Ethiopia] and ICF. Mini Ethiopia Demographic and Health Survey 2019: Key Indicators Report. Addis Ababa, Ethiopia, and Rockville, Maryland, USA. CSA and ICF. 2019.
- [Derived] Yoseph A, Teklesilasie W, Guillen-Grima F, Astatkie A. Effect of community health education on mothers' knowledge of obstetric danger signs and birth preparedness and complication readiness practices in southern Ethiopia: A cluster randomized controlled trial. PLoS One. 2024 Nov 27;19(11):e0312267. doi: 10.1371/journal.pone.0312267. eCollection 2024. PMID 39602439
- [Derived] Yoseph A, Teklesilasie W, Guillen-Grima F, Astatkie A. Community-Based Health Education Led by Women's Groups Significantly Improved Maternal Health Service Utilization in Southern Ethiopia: A Cluster Randomized Controlled Trial. Healthcare (Basel). 2024 May 18;12(10):1045. doi: 10.3390/healthcare12101045. PMID 38786455